CLINICAL TRIAL: NCT00619008
Title: Energy and Appetite Regulation by High and Low CHO Diets
Brief Title: Energy Balance Weight Regulation Study
Acronym: BALANCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Diane D. Stadler, Oregon Health & Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R21AT002753 (NIH)
Record Dates: First submitted 2008-02-15; First posted 2008-02-20 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
Keywords: obesity; low carbohydrate diet; high complex carbohydrate diet; weight regulation hormones; hunger; satiety; energy expenditure; body composition; weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Ad libitum low carbohydrate diet
  Interventions: Other: Ad libitum low carbohydrate diet
- 2 (Experimental): Ad libitum high complex carbohydrate diet
  Interventions: Other: Ad libitum High Complex Carbohydrate Diet
- 3 (Experimental): Energy-restricted high complex carbohydrate diet
  Interventions: Other: Energy-restricted high complex carbohydrate diet

INTERVENTIONS:
Other: Ad libitum low carbohydrate diet — 6 week ad libitum low carbohydrate diet
  Other Names: Low Carb diet
  Arms: 1
Other: Ad libitum High Complex Carbohydrate Diet — 6 week ad libitum high complex carbohydrate diet
  Other Names: DASH diet
  Arms: 2
Other: Energy-restricted high complex carbohydrate diet — 6 week energy-restricted (68% of estimated energy requirement for weight maintenance) high complex carbohydrate diet.
  Other Names: Energy-restricted DASH diet
  Arms: 3

SUMMARY:
The purpose of this study is to test the hypothesis that a low-carbohydrate diet will impact hormones and other factors that regulate appetite and energy balance, and result in lower energy intake and greater weight loss, than a high complex carbohydrate diet.

DETAILED DESCRIPTION:
The rising epidemic of obesity in the United States is accompanied by widespread public use of low carbohydrate diets for weight loss. The popularity of these diets is due partly to the promise of a "metabolic advantage" that promotes faster weight loss without an overriding sense of hunger. If this claim is true, we hypothesize that a low-carbohydrate diet will impact hormones and other factors that regulate appetite and energy balance, and result in lower energy intake and greater weight loss, than a high complex carbohydrate diet. To test this hypothesis, we will conduct a randomized, controlled feeding trial in which obese adults will be randomly assigned to one of three interventions: a low-carbohydrate-ad libitum diet, a high-carbohydrate-ad libitum diet, or a high-carbohydrate-energy-restricted diet. The low-carbohydrate diet will be modeled after the Induction Phase of the Atkins Diet. The high carbohydrate diet will be based on the "Dietary Approaches to Stop Hypertension (DASH)" diet. Participants will eat a standardized weight maintenance diet for 3 weeks. Then, for 6-weeks, participants assigned to either ad libitum group will be given their assigned diet at 120% of there estimated energy needs to maintain weight and allowed to eat as much as desired. Participants assigned to the energy-restricted group will be provided a DASH diet at 67% of their estimated energy needs to maintain weight and asked to eat all foods provided. Food intake will be measured daily. Body weight and hunger and satiety scores will be measured three times a week. Body composition and energy expenditure will be measured before and after the intervention. 24-hour profiles of hormones and other factors that influence central appetite and weight regulation (insulin, leptin, ghrelin, PYY, GLP-1) will be measured before, and on first and last days of the intervention, to compare acute and chronic metabolic effects of the diets. The analysis of primary outcomes will be based on repeated measures and longitudinal models methodology. This study offers a unique opportunity to explore how extreme differences in dietary composition, before and after weight loss, affect components of energy balance and markers of central appetite and weight regulation. These results will be used to design hypothesis-driven studies of the identified mediators of appetite and weight regulation in response to dietary manipulation.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-50 kg/m2
* Age 21-65 years
* Relative good health

Exclusion Criteria:

* Major debilitating mental of physical illness that would interfere with participation
* Renal or hepatic disease, diabetes, gallbladder disease, untreated hyper-or hypothyroidism, poorly controlled hypertension (>3 HT medications)
* Use of lipid lowering medications
* Current of recent (within 12 mo) pregnancy or lactation
* Current excessive use of alcohol
* Current/recent (within 1 year)use of tobacco products
* Food allergies, food restrictions, or food preferences that are inconsistent with the research diets

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
24-hour profiles and AUCs of hormones and other factors that influence central appetite and weight regulation (insulin, leptin, ghrelin, PYY, GLP-1). | Week 2, week 3 and week 9 of intervention

SECONDARY OUTCOMES:
Energy intake, hunger and satiety ratings | week 2, 3, and 9 of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Diane D Stadler, PhD, Principal Investigator — OSHU
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States